CLINICAL TRIAL: NCT02202603
Title: A Three Stage, Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Oral PTH (1-34) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entera Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0020-11-HMO-EnteraBio
Record Dates: First submitted 2011-06-20; First posted 2014-07-29 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Drug Safety
MeSH Terms: interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Teriparatide group 1 (Active Comparator): Subcutaneous injection of Teriparatide
  Interventions: Drug: Teriparatide
- excipients (Placebo Comparator): Oral pill without API
  Interventions: Drug: placebo
- API (Experimental): Oral administration of pill with API
  Interventions: Drug: Teriparatide
- API optimization 1 (Experimental): Oral administration of pill with API, for PK optimization #1
  Interventions: Drug: Teriparatide
- API optimization 2 (Experimental): Oral administration of pill with API, for PK optimization #2
  Interventions: Drug: Teriparatide
- API optimization 3 (Experimental): Oral administration of pill with API, for PK optimization #3
  Interventions: Drug: Teriparatide
- API optimization 4 (Experimental): Oral administration of pill with API, for PK optimization #4
  Interventions: Drug: Teriparatide
- API optimization 5 (Experimental): Oral administration of pill with API, for PK optimization #5
  Interventions: Drug: Teriparatide
- API optimization 6 (Experimental): Oral administration of pill with API, for PK optimization #6
  Interventions: Drug: Teriparatide
- API optimization 7 (Experimental): Oral administration of pill with API, for PK optimization #7
  Interventions: Drug: Teriparatide
- Teriparatide group 2 (Active Comparator): Subcutaneous injection of Teriparatide
  Interventions: Drug: Teriparatide
- Excipients (Experimental): Oral pill without API
  Interventions: Drug: placebo
- API Optimized (Experimental): expanded group size with API in optimized dosage and administration form.
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — single oral tablet
  Arms: API; API Optimized; API optimization 1; API optimization 2; API optimization 3; API optimization 4; API optimization 5; API optimization 6; API optimization 7
Drug: Teriparatide — subcutaneous standard injection
  Arms: Teriparatide group 1; Teriparatide group 2
Drug: placebo — Oral placebo
  Arms: Excipients; excipients

SUMMARY:
A Double blinded (oral), Open Label, Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Oral PTH (1-34) in healthy Subjects to establish the safety, tolerability, bioavailability, pharmacokinetic, and pharmacodynamic profile and the of Entera's oral PTH(1 - 34) in adult healthy human volunteers.

DETAILED DESCRIPTION:
This study will have three stages. Stage 1: Safety and initial bioavailability of Entera's oral EP101 in adult male healthy volunteers. (SA-BA) Stage 2: Assessment of bioavailability and safety of Entera's oral EP101 in adult male healthy volunteers. (SA-BA-PK-PD) Stage 3: Safety, PK, and PD of final dose of Entera's oral PTH(1 - 34) in adult healthy male and female volunteers. (SA-BA-PK-PD)

ELIGIBILITY:
Inclusion Criteria:

* ● Signed Informed consent to the study.

  * Male and female volunteers ,aged 18 - 50 years, BMI 18-30 kg/m2, inclusive,
  * Subjects able to adhere to the visit schedule and protocol requirements
  * Hematology ,Chemistry and Urinalysis values with no clinical significance or do not reflect a medical condition which according to the physicians' judgment might confound the results of the study or pose additional risk to the subject by participation in the study.
  * Hemoglobin level >. 12.5 g/dl
  * Blood pressure levels with no clinical significance.
  * Negative serology to HIV, Hepatitis B, Hepatitis C.
  * No known drug and alcohol abuse
  * Negative urinary drugs of abuse at screening
  * No allergy to soy bean products.
  * No prescription medications taken within one month to enrollment
  * Over-the-counter drugs (including vitamins) taken within 14 days prior to visit 2 are subject to the investigators' discretion for inclusion.
  * No subjects with previous urolithiasis.
  * Non-smoking,
  * In good health as determined by past medical history, physical examination, vital signs, electrocardiogram and laboratory tests at screening

Exclusion Criteria:

* ● Concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.

  * Treatment with any investigational product within the last 30 days, enrollment or intention to enroll in any active study involving the use of investigational devices or drugs.
  * Presence of any other condition or circumstance that, in the judgment of the Investigator, might increase the risk to the patient or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
  * Active infections
  * History of drug or alcohol abuse
  * Known allergies or sensitivities to components of study treatment or study procedures, including Soy.
  * Clinically diagnosed psychiatric disorders that may interfere with patient study participation
  * Medical history known or suspected to increase risks of AEs related to study drug, up to the investigator's discretion
  * Chronic illnesses, up to the investigator's discretion
  * Female subjects must have a negative serum pregnancy test at screening and be willing and able to use a medically acceptable method of birth control (non-hormonal intrauterine device with condom, or diaphragm with condom, or condom with spermicide) from the screening visit through the study termination visit or declare that they are abstaining from sexual intercourse from the screening visit through the study termination visit or are surgically sterile (have undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or post menopausal. Postmenopausal women are defined as women with menstruation cessation for 12 consecutive months prior to signing of the informed consent form.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to 17 weeks
  throughout the study beginning from the time the subject signs the consent form until the end of study, subjects will complete the following evaluations:
  * Vital signs (blood pressure, heart rate, oral temperature)
  * Clinical laboratory evaluations, hematology, chemistry
  * Physical Exam
  * ECG

CONTACTS AND LOCATIONS:
Overall Officials: Yosef Caraco, MD, Principal Investigator — Hadassah Ein Kerem Medical Center
Locations (1):
- HMO Clinical Research Center Hadassah Ein Kerem Medical Center, Jerusalem, Israel